CLINICAL TRIAL: NCT04740710
Title: Breathing and Attention Training for Chronic Low Back Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Breathe for Pain; OCR39823 (Other: UF OnCore); IRB202002612 (Other: UF IRB-01)
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic Pain; Low Back Pain; Breathing
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Respiratory Aspiration | interventions — Respiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Breathing and Attention Training (Active Comparator): The standard breathing and attention training (BAT) includes guided instructions on deep breathing and relaxation. Participants will practice standard BAT once a day for 15 minutes for 5 days in a row.
  Interventions: Behavioral: Breathing and Attention Training
- Focused Breathing and Attention Training (Experimental): The focused BAT is similar to the standard BAT in most ways but includes extra instructions to help focus and alter breathing patterns. Participants will practice focused BAT once a day for 15 minutes for 5 days in a row.
  Interventions: Behavioral: Breathing and Attention Training

INTERVENTIONS:
Behavioral: Breathing and Attention Training — A guided audio recording will instruct participants to alter their breathing and pay attention in specific ways.

SUMMARY:
The purpose of this research study is to see if breathing and attention training (BAT) treatments improve pain symptoms and well-being in people who have chronic low back pain (cLBP). For this breathing intervention, you will be randomly assigned to either standard or focused BAT. The standard BAT includes instructions on deep breathing and relaxation. The focused BAT is similar to the standard BAT in most ways but includes extra instructions to help you focus and alter your breathing patterns.

DETAILED DESCRIPTION:
The primary objective of the proposed pilot randomized controlled trial (RCT) is to examine the safety, feasibility, and acceptability of a 5-day breathing and attention training (BAT) in a sample of 30 adults with cLBP. The secondary objective is to explore preliminary clinical efficacy and potential mechanisms of the breathing interventions (focused-BAT and standard-BAT), by examining changes in clinical pain outcomes and potential pain-related psychological, physiological, and behavioral mediating variables. Both interventions will be delivered via an audio recording in order to standardize the interventions across participants and to enhance treatment fidelity. Results from this study will inform the successful design and implementation of a larger RCT and provide preliminary evidence regarding the potential efficacy of this breathing intervention for people with cLBP.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain consistent with recommendations of the NIH task force on cLBP (i.e., participants with cLBP of at least moderate impact that has persisted on more days than not over the past 3 months)
* Age 18-65

Exclusion Criteria:

* Systemic rheumatic disease/condition (e.g. rheumatoid arthritis, systemic lupus erythematosus, fibromyalgia).
* Asthma, breathing problems, or a respiratory disorder (e.g., chronic obstructive pulmonary disease).
* Daily use of opioids. We will exclude patients using opioids daily as both continued use and temporary withdrawal from these medications this could affect pain perception and response to interventions. Other medications being used will be recorded and controlled in statistical analyses as needed.
* Uncontrolled hypertension (i.e. SBP/DBP of > 150/95), orthostatic hypotension, cardiovascular or peripheral arterial disease. These exclusions are in place primarily for safety reasons, however, uncontrolled hypertension can also affect pain perception, which is another reason for excluding these individuals.
* Neurological disease (e.g. Parkinson's, multiple sclerosis, epilepsy, vasovagal syncope) or evidence of previous brain injury, including stroke and traumatic brain injury.
* Serious psychiatric disorder requiring hospitalization within the past 12 months or characterized by active suicidal ideation.
* Current substance use disorder or history of hospitalization for treatment of substance use disorder.
* Pregnant
* Any significant comorbidities that, in the opinion of the investigators, could interfere with the study or lead to deleterious effects for the patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-07-18 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Treatment Satisfaction Questionnaire | 3-months
  Treatment acceptability and participant satisfaction will be measured with several items rated on a 10-point scale where higher scores represent greater treatment acceptability and satisfaction.
Incidence of Adverse Events | Through study completion, up to 3-months
  Number of serious adverse events

SECONDARY OUTCOMES:
Change in Pain Intensity | Baseline, Day 1, Day 2, Day 3, Day 4, Day 5
  Numerical rating scale (1- "No pain", 10- "Worst pain imaginable") of current pain intensity measured before and after each intervention session.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared upon request by other researchers.

REFERENCES:
- [Derived] Pratscher SD, Sibille KT, Fillingim RB. Conscious connected breathing with breath retention intervention in adults with chronic low back pain: protocol for a randomized controlled pilot study. Pilot Feasibility Stud. 2023 Jan 24;9(1):15. doi: 10.1186/s40814-023-01247-9. PMID 36694217